CLINICAL TRIAL: NCT01755715
Title: Immediate Versus Later Insertion of IUD After Medical Termination of Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riina Korjamo (Other)
Responsible Party: Sponsor-Investigator, Riina Korjamo, MD, Helsinki University Central Hospital
Organization: Helsinki University Central Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KILKE
Record Dates: First submitted 2012-12-13; First posted 2012-12-24 (Estimated); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Contraception After Medical Abortion
Keywords: Abortion; Contraception; Intrauterine Devices; Intrauterine Device Expulsion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): Insertion of IUD at 2-4 weeks after abortion.
- Immediate IUD insertion (Experimental): Insertion of IUD immediately (at the same day to 3 days) after expulsion of placenta.
  Interventions: Procedure: Immediate IUD insertion

INTERVENTIONS:
Procedure: Immediate IUD insertion — Insertion of LNG-IUD (Mirena) (at the same day to 3 days) after expulsion of placenta.
  Arms: Immediate IUD insertion

SUMMARY:
The main objective of this study is to compare, in a randomised, controlled and prospective fashion, initiation of intrauterine contraception (IUC) at about immediate (0 to 3 days) versus 2 to 4 weeks post medical abortion with regard to expulsions and use of contraception one year after abortion.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Planning medical abortion
* Planning LNG-IUD (Mirena) contraception

Exclusion Criteria:

* Pathological pregnancies or abnormality of the uterus or cervix
* Acute endometritis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2013-01; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Number of expulsions | 1 year
  Number of IUD expulsions
Use of IUD | 1 year

SECONDARY OUTCOMES:
Bleeding profile | 3 months
Repeat abortions | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Oskari Heikinheimo, MD, PhD, Study Director — Helsinki University Central Hospital; Maarit Mentula, MD, PhD, Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Helsinki University Central Hospital, Dept Ob&Gyn, Helsinki, Finland